CLINICAL TRIAL: NCT01038466
Title: Follow-Up Observational Study In CHAT Trial Participants With Advanced And/Or Metastatic Breast Cancers That Overexpress HER2, Who Were Randomised To Receive Trastuzumab And Docetaxel With Or Without Capecitabine
Brief Title: Observation Only Study Involving Participants Enrolled in the CHAT Trial
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Contact Asia Pacific (Network)
Responsible Party: Associate Professor Richard Bell, Contact Asia Pacific
Other Study IDs: CB.0901
Record Dates: First submitted 2009-09-10; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-09

CONDITIONS: Breast Cancer
Keywords: CHAT; breast cancer; non interventional observational study
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CHAT trial participants: CHAT trial participants whose data was used in the final data analysis for the CHAT study

SUMMARY:
The aim of the CHAT study ("An open-label, randomized Phase II study of Herceptin (trastuzumab), Taxotere® (docetaxel) and Xeloda (capecitabine) in combination, versus Herceptin (trastuzumab) plus Taxotere® (docetaxel), in patients with advanced and/or metastatic breast cancers that overexpress HER2") was to test the combination of Trastuzumab and Docetaxel with or without capecitabine as first-line therapy for HER2 positive locally advanced or metastatic breast cancer.

Overall Response Rate was the primary endpoint of the CHAT study. This study failed to meet its primary objective of showing a difference between the treatment groups, with equivalent high response rates for the Trastuzumab plus Docetaxel and Trastuzumab, Docetaxel plus capecitabine arms.

Secondary endpoints in the CHAT study were Progression-Free-Survival, Time-to-Progression, Overall Survival, duration of response and safety profile. Whilst analysis of the existing data is consistent with improvement with the triplet therapy, interpretation is compromised by the relatively short median follow-up of 24 months. In hindsight the statistical design was flawed by selection of a sub optimal primary endpoint and consequently data was collected and analysed early in relation to time-dependent endpoints. Beyond CHAT will permit capture of mature data for time-related endpoints. Time-to-Progression and Overall Survival are the co-primary endpoints for the Beyond CHAT protocol. The impact of treatment following the first progression, on survival, will be explored.

Time-to-Progression will be defined from the time interval between the date of randomisation and the occurrence of progressive disease under therapy according to RECIST criteria.

Overall Survival will be defined as the time from date of randomisation to date of death

DETAILED DESCRIPTION:
The objective of this study is to gain mature data on the long-term efficacy of the combination of Trastuzumab and Docetaxel with or without capecitabine as first-line therapy for HER2 positive locally advanced or metastatic breast cancer.

The study also aims to gain information on the additional treatments and sequencing used in patients that have progressed following the combination of Trastuzumab and Docetaxel with or without capecitabine as first-line therapy for HER2 positive locally advanced or metastatic breast cancer.

Overall Survival data on patients who have progressed following the combination of Trastuzumab and Docetaxel with or without capecitabine as first-line therapy for HER2 positive locally advanced or metastatic breast cancer will also be analysed and reported.

ELIGIBILITY:
Inclusion Criteria:

* CHAT trial participants whose data was used in the final data analysis for the CHAT study

Exclusion Criteria:

* Any patients who have withdrawn consent to the CHAT study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All 222 CHAT trial participants whose data was used in the final data analysis for the CHAT study will be included in the Beyond CHAT follow-up observational study
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
The primary endpoints are Time-to-Progression and Overall Survival in the two treatment arms of the CHAT study. | survival

SECONDARY OUTCOMES:
Progression-Free-Survival | 7 years
Overall Survival | 7 years
Anatomical sites of progression | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bell, MBBS, Principal Investigator — Contact Asia Pacific
Locations (1):
- CONTACT Asia Pacific, Geelong, Victoria, Australia